CLINICAL TRIAL: NCT04995848
Title: Elepalliation - Digital Platform for Patienter i Palliation og Deres pårørende
Brief Title: Telepalliation - Digital Platform for Patients in Palliation and Their Relatives
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University (Other)
Collaborators: Palliative Team,Hospital of South West Jutland (Unknown); Center for Innovative Medical Technologies (CIMT), Odense University Hospital (Unknown); Danish Cancer Society (Other); Laboratory of Welfare Technology, Department of Health Science and Technology, Aalborg University (Unknown)
Responsible Party: Principal Investigator, Birthe Dinesen, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: N-20200094
Record Dates: First submitted 2021-05-26; First posted 2021-08-09 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Heart Failure; Chronic Obstructive Pulmonary Disease; Neurological Diseases
Keywords: Palliative care; Palliation; Platform; Quality of life
MeSH Terms: conditions — Neoplasms; Heart Failure; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: Mixed method randomised control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telepalliation group (Experimental): The intervention group will participate in the telepalliation program. The patients will lent a tablet during the RCT study to access the TelePal.dk platform an video consultations. The patients will participate from the time they are referred to palliative care, and are enrolled in the telepalliation program for up to six months or until:
  1. They stop being followed by the Palliative Team due to lack of symptoms
  2. They are diagnosed with delirium based upon clinical guidelines and the Confusion Assessment Method (CAM). The assessment of delirium will be done by either:
     * The project nurse or the clinical responsible doctor at the patients' home OR
     * A district nurse under video supervision by the project nurse or the clinical responsible doctor
  3. Death of the patient
  Interventions: Other: Telepalliation
- Conventional palliation program (No Intervention): The control group will follow a conventional palliation program. The patients will participate from the time they are referred to palliative care, and are enrolled in the telepalliation program for up to six months or until:
  1. They stop being followed by the Palliative Team due to lack of symptoms
  2. They are diagnosed with delirium based upon clinical guidelines and the Confusion Assessment Method (CAM). The assessment of delirium will be done by either:
     * The project nurse or the clinical responsible doctor at the patients' home OR
     * A district nurse under video supervision by the project nurse or the clinical responsible doctor
  3. Death of the patient

INTERVENTIONS:
Other: Telepalliation — Telepalliation platform Telepal.dk
  Arms: Telepalliation group

SUMMARY:
This project has focus on patients in palliation testing a digital platform TelePal.dk.

DETAILED DESCRIPTION:
The aim of the RCT study is to:

• Test, implement, and evaluate a telepalliation program for patients receiving palliative care (cancer, heart failure (HF), COPD, and motor neuron disease) from a clinical, psychosocial, inter-organizational, and health economic perspective.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years
* Live in Esbjerg, Varde, Billund, Fanø or Vejen Municipality
* Cancer, heart failure, chronic obstructive pulmonary disease (COPD), and motor neuron disease (neurological diseases) referred to the Palliation Team at Southwest Jutland Hospital
* Basic computer skills or a relative who has basic computer skills

Exclusion Criteria:

* Delirium at enrolment based on CAM score
* Active psychiatric history (as noted in the medical record) other than depression or anxiety related to the main diagnosis referred to palliative care
* Lack of ability to cooperate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Quality of life | At baseline, week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
  Measured by the European Organization for Research and Treatment of Cancer, questionnaire regarding quality of life in palliative cancer care patients (EORTC QLQ-C15-PAL).

SECONDARY OUTCOMES:
Changes in medicine | At enrolment and week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
  Information on medicine for both groups will be collected at enrolment and every week from the electronic patient record (EPR). Changes in medicine over time will be analyzed.
Changes in feeling of security | At baseline, twice every week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
  Measured on a likert scale
Experiences of pain | At baseline, week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
  Numerical Rating Scale (NRS)
Experience of pain (brief) | At baseline, week 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26
  Brief Pain Inventory, short form (BPI-sf)
Experiences of patients on the actual use of the TelePal.dk platform and their experiences of being a part of a telepalliation program | Week 4
  Qualitative interviews
Experiences of relatives on the actual use of the TelePal.dk platform and their experiences of being a part of a telepalliation program | Week 4 and 3 months
  Qualitative interviews
Experiences of health care professionals on the actual use of the TelePal.dk platform and their experiences of being a part of a telepalliation program | 6 months and 12 months
  Qualitative interviews
Perceptions on usability of a cross-sector communication platform and telerehabilitation program by patients, relatives and health care professionals | 12 months
  Qualitative interviews
Observations on usability of a cross-sector communication platform and telerehabilitation program by patients, relatives and health care professionals | 12 months
  Observations
Health related quality of life | week 1 and week 4
  Measured by EQ-5D Health Questionnaire
Cost of healthcare services | 24 months
  Cost-effectiveness analysis ((number of phone/video calls, equipment, driving, personal use in palliative care (video and home visits), visits to general practitioner and outpatient clinic, hospitalizations, readmissions and length of stay, visits from palliative team))

CONTACTS AND LOCATIONS:
Overall Officials: Birthe Dinesen, MSc, PhD, Principal Investigator — Aalborg University; Jarl Voss Andersen Sigaard, MD, Study Director — Palliative Team, South West Jutland Hospital
Locations (1):
- Palliative Team, South West Jutland Hospital, Esbjerg, Denmark

IPD SHARING:
Plan to Share IPD: No
No plan for sharing protocol as we are applying for patent.

REFERENCES:
- [Derived] Sigaard JVA, Joensen EDR, Birgisdottir UR, Spindler H, Dinesen B. Telepalliation creates a sense of security: A qualitative study of patients with cancer receiving palliative care. Palliat Med. 2025 Oct 7:2692163251364145. doi: 10.1177/02692163251364145. Online ahead of print. PMID 41055129
- [Derived] Sigaard JVA, Henneberg NC, Schacksen CS, Kronborg SH, Petrini L, Kidholm K, Birgisdottir UR, Spindler H, Dinesen B. A Digital Platform (Telepalliation) for Patients in Palliative Care and Their Relatives: Protocol for a Multimethod Randomized Controlled Trial. JMIR Res Protoc. 2024 Apr 2;13:e49946. doi: 10.2196/49946. PMID 38564264
- See also: Read more about the Laboratory for Welfare Technology - telehealth and telerehabilitation, Aalborg University — http://www.labwelfaretech.com/en/